CLINICAL TRIAL: NCT02064465
Title: A Single-Dose, Open-Label, Randomized, Parallel-Group Study to Demonstrate the Bioequivalence of Lamotrigine Dispersible/Chewable Tablet (100mg) and Lamotrigine Compressed Tablet (100mg) in Healthy Chinese Male Subjects
Brief Title: The Bioequivalence Study of Lamotrigine Dispersible/Chewable Tablets 100mg Compared With Compressed Tablet 100 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200697
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamotrigine Dispersable/Chewable (Experimental): lamotrigine dispersible/chewable tablet 100mg
  Interventions: Drug: Lamotrigine Dispersible/Chewable tablet
- Lamotrigine Compressed (Experimental): lamotrigine compressed tablet 100mg
  Interventions: Drug: Lamotrigine Compressed tablet

INTERVENTIONS:
Drug: Lamotrigine Dispersible/Chewable tablet — Single dose of lamotrigine dispersible/chewable 100mg tablet at Day1
  Other Names: Lamictal
  Arms: Lamotrigine Dispersable/Chewable
Drug: Lamotrigine Compressed tablet — Single dose of lamotrigine compressed 100mg tablet at Day1
  Other Names: Lamictal
  Arms: Lamotrigine Compressed

SUMMARY:
This is an open-label, randomised, parallel-group study to demonstrate the bioequivalence of lamotrigine 100mg in two different formulations, dispersible/chewable tablet and compressed tablet, in healthy subjects under fasting conditions. Subjects will be randomized in equal numbers to be dosed with either lamotrigine dispersible/chewable (Test) 100mg tablet or lamotrigine compressed (Reference) 100mg tablet. Pharmacokinetic blood sampling will be collected over 216 hours post dose. Safety (tolerability) will be observed up to 216 hours post dose. Safety assessments will include regular monitoring of vital signs, ECG's, adverse events (AEs) and safety laboratory tests. A follow-up visit is scheduled within 10-17 days post-dose.

DETAILED DESCRIPTION:
This is a single dose, open-label, randomized, parallel-group study to demonstrate the bioequivalence of lamotrigine dispersible/chewable tablet and lamotrigine compressed tablet at 100mg in healthy Chinese male subjects in fasting conditions. Approximate 138 Chinese healthy male subjects will be enrolled in accordance with the inclusion and exclusion criteria. Subjects will be 18 to 45 years, healthy and body mass index between 19-24 kg/m2 and sign the informed consent.

Having given written informed consent, subjects will be required to undergo a pre-study medical screen within 14 days of the dosing day. Subjects will be admitted on Day 0 (the day before dosing) and will stay in the unit until after the 24-hour post-dose assessments on Day 2. The time that a subject is discharged from the unit may be agreed with unit staff but subjects must return for all designated pharmacokinetic (PK) samples and on scheduled time for observation.

The subjects will be randomized in equal numbers to be dosed under fasting conditions with either lamotrigine dispersible/chewable tablet or lamotrigine compressed tablet. The pharmacokinetic assessment will last 10 days. The blood samples will be collected immediately before dosing (pre-dose) and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168 and 216 hours post dose for determination of lamotrigine concentration in blood. Safety and tolerability evaluation will be observed up to 216 hours post-dose, including adverse events, vital signs, physical examination, electrocardiogram. All subjects will be required to undergo a follow-up assessment within 10-17 days after receiving the study medication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male non-smoker, based on medical history and physical examination, aged between 18 and 45 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator (in consultation with the GlaxoSmithKline (GSK) Medical Monitor if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kg and BMI within the range 19 - 24 kg/m2 (inclusive).
* Capable of returning to study site for follow-up according to the requirement of protocol and willing to comply with the policy, procedure and restriction of the study.
* Capable of reading and understanding the information listed in the consent form. Signing the informed consent prior to any study related procedure.
* Aspartate transaminase (AST), Alanine transaminase (ALT), alkaline phosphatase (ALP) and total bilirubin <= 1.5✕Upper limit of normal (ULN) (total bilirubin >1.5 x ULN alone is acceptable if direct bilirubin <35% of total bilirubin).
* Normal blood pressure (systolic blood pressure 90-140 mmHg, inclusive, diastolic blood pressure < 90mmHg) and pulse rate (60-100, inclusive).
* No clinically significant abnormality on 12-lead ECG.
* Corrected QT interval (QTc) < 450 ms; or corrected QT interval < 480 ms for subjects with bundle-branch block, based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period.
* Male subjects with female partners of child-bearing potential must use one of the contraceptive methods after the first dose of study treatment and until the follow-up visit.

Exclusion Criteria:

* Current or chronic history of cardiovascular, respiratory, gastrointestinal, endocrine, hematological, psychical or nervous system diseases, use of drug that can change the absorption, metabolism or elimination of study drug, or result in danger or other drugs or diseases that interfere with the interpretation of study data.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities or Gilbert's syndrome (with the exception of asymptomatic gallstones).
* Current or past history of nervous-psychiatric disorder, as assessed by Columbia Suicide Severity Rating Scale-baseline evaluation or in the opinion of investigator that the subject is at risk of suicide or with history of suicide behavior/attempt.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* Consumption of grapefruit or grapefruit juice within 7 days prior to first dose of study medication.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of asthma, anaphylaxis or anaphylactic reactions, severe allergic responses.
* Subjects who have received lamotrigine previously (subjects who received placebo in a previous study will be allowed)
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days prior to the dosing day, which in the opinion of the Principal Investigator, may interfere with the study procedures or compromise safety.
* A positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody (HCAb) result at screening
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody at screening.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2014-03-15 (Actual); Primary Completion 2014-07-08 (Actual); Study Completion 2014-07-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve [AUC(0-inf)] of lamotrigine if coefficients of variation (CV)% of λz<=30%, or AUC(0-inf)• λz if CV% of λz >30%, or AUC(0-t) if AUC(0-inf) cannot be accurately determined, including bioequivalence evaluation | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 216 hours post-dose
The observed maximum serum drug concentration (Cmax), including bioequivalence evaluation | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 216 hours post-dose

SECONDARY OUTCOMES:
Time to reach Cmax (Tmax) as data permit. | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 216 hours post-dose
Elimination half-time (t1/2) as data permit | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 216 hours post-dose
Elimination rate constant, linear regression according to linear serum drug concentration-time curve (λz) as data permit. | pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 216 hours post-dose
Safety and tolerability as measured by adverse events, vital sign, ECG and clinical laboratory measurements. | at screeing, Day0-10, follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 200697 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200697?search=study&study_ids=200697#rs
- Available data/document: Statistical Analysis Plan: 200697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200697 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register